CLINICAL TRIAL: NCT04172844
Title: A Multisite Phase Ib Study of Pevonedistat, Azacitidine (or Decitabine), and Venetoclax (PAVE) for the Treatment of Patients With Acute Myelogenous Leukemia (AML)
Brief Title: Pevonedistat, Azacitidine (or Decitabine), and Venetoclax for the Treatment of Patients With Acute Myelogenous Leukemia
Acronym: PAVE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Takeda P3001 study didn't meet primary endpoint of improvement in event-free survival. There is no regulatory path forward for pevonedistat.
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Ehab L Atallah, Professor, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRO36496
Record Dates: First submitted 2019-11-20; First posted 2019-11-21 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Acute Myelogenous Leukemia
Keywords: leukemia; acute myeloid leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — Azacitidine; venetoclax; pevonedistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pevonedistat Dose Escalation (Experimental): This study uses a varied 3 + 3 design. Three patients will be started at a dose of 10 mg/m^2 days 1, 3 and 5. If no DLTs are observed in the first 3 participants, then a new cohort will be enrolled at the next planned dose level of 15 mg/m^2 days 1, 3 and 5. If two out of three subjects experience a DLT, then they will de-escalate one dose level. If one subject in three experiences a DLT, then expand up to three subjects at 20 mg/m^2 day 1, 3 and 5. If two out of six subjects experience a DLT, de-escalate one level. All subjects will receive Azacitidine and Venetoclax at the indicated dosages and timing.
  Interventions: Drug: Azacitidine; Drug: Venetoclax; Drug: Pevonedistat
- Dose Expansion Phase (Experimental): Patients will receive the recommended phase 2 dose (RP2D) identified from dose-escalation phase.
  Interventions: Drug: Azacitidine; Drug: Venetoclax; Drug: Pevonedistat

INTERVENTIONS:
Drug: Azacitidine — 75mg/m^2 Days 1-7 given IV
  Other Names: 5 AZC; 5-AC; 5-Azacytidine; 5-AZC; Azacytidine; Azacytidine, 5-; Ladakamycin; Mylosar; U-18496; Vidaza
Drug: Venetoclax — 100 mg on cycle 1 day 1, 200 mg daily on cycle 1 day 2, 400 mg on cycle 1 day 3 and thereafter from cycle 1. Venetoclax is given for a minimum of 21 days and a maximum of 28 days. Administered orally.
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto
Drug: Pevonedistat — The doses for the 3 + 3 design (dose escalation phase) are listed in the arm description. The dose-expansion phase will use the maximum-tolerated dose.
  Other Names: MLN4924; Nedd8-Activating Enzyme Inhibitor MLN4924

SUMMARY:
This is a phase Ib study with a 3 + 3 dose escalation design followed by a dose-expansion phase.

DETAILED DESCRIPTION:
The study hypothesis is that the combination of pevonedistat, azacitidine, and venetoclax will be effective, safe, and well tolerated in patients with AML.

The primary objective of this portion of the study is to determine a recommended phase 2 dose (RP2D) of pevonedistat, azacitidine, and venetoclax. The investigators will use a variation of the 3+3 design where both escalation and de-escalation are possible. A minimum of nine and a maximum of 24 subjects will be needed for the phase 1 part of the study (dose-escalation phase). The dose limiting toxicity (DLT) observation period for dose escalation will be during cycle 1.

Prior to enrolling patients at the next applicable dose level, all patients must complete the DLT period of the current dose level. The Data Safety Monitoring Committee will review the results of each dose level before the next applicable dose level opens for enrollment.

Dose Expansion Phase

The primary objective of this portion of the study is to confirm the feasibility and tolerance of the combination of pevonedistat, azacitidine, and venetoclax in patients with AML. Given that the dose-escalation phase described above will be able to establish the RP2D, the dose-expansion phase will employ this dose. In addition to relapsed/refractory AML patients, newly diagnosed AML patients can also be included in this phase to assess the feasibility and tolerance of this combination regimen.

A minimum of six patients will be enrolled in the dose-expansion phase, which could be expanded based on the safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Male or female subjects 18 years or older.
* Patients must have a diagnosis of morphologically documented AML or secondary AML [from prior conditions, such as myelodysplastic syndrome (MDS), or therapy-related AML (t-AML), as defined by World Health Organization (WHO) criteria.
* During the dose-escalation phase, only subjects with relapsed/refractory AML will be eligible.
* During the expansion phase, subjects with relapsed/refractory AML will be eligible OR subjects with newly diagnosed AML unable or unwilling to receive intensive induction chemotherapy will be eligible.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Clinical laboratory values within the following parameters:
* Albumin >2.7 g/dL.
* Total bilirubin ≤ institutional upper limit of normal (ULN). Patient with total bilirubin > ULN may enroll if direct bilirubin ≤1.5 x institutional ULN of the direct bilirubin.
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × institutional ULN.
* Creatinine clearance ≥ 30 mL/min (calculated by Cockcroft-Gault formula).
* White blood cell (WBC) count < 25,000/μL before administration of pevonedistat on cycle 1 day 1. (Note: Hydroxyurea may be used to meet this criterion.)
* Prothrombin time (PT) and partial thromboplastin time (PTT) < 1.5 institutional ULN.
* Female subjects who:
* Are postmenopausal for at least one year before the screening visit, OR
* Are surgically sterile, OR
* If they are of childbearing potential:
* Agree to practice one highly effective method and one additional effective (barrier) method of contraception, at the same time, from the time of signing the informed consent through four months after the last dose of study drug (female and male condoms should not be used together), OR
* Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception).
* Male subjects, even if surgically sterilized (i.e., status postvasectomy), who:
* Agree to practice effective barrier contraception during the entire study treatment period from the time of signing the informed consent through and through four months after the last dose of study drug (female and male condoms should not be used together), OR
* Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods for the female partner] withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.)

Exclusion Criteria:

* Acute promyelocytic leukemia.
* Extramedullary only relapse AML.
* Treatment with systemic antineoplastic therapy or radiation within 14 days before the study enrollment. The use of hydroxyurea for leukoreduction is permitted. Subjects must have recovered from the side effects of prior therapy per treating physician discretion.
* Hematopoietic Stem Cell Transplantation (HCT) within 100 days of enrollment, or evidence of veno-occlusive disease (VOD) at any time post-transplant, or active acute graft-versus-host disease requiring systemic immunosuppressive therapy.
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of study procedures.
* Current systemic treatment with strong or moderate cytochrome P3A (CYP3A) inducers within seven days prior to enrollment.
* Any evidence of spontaneous tumor lysis syndrome (TLS).
* Active, significant, uncontrolled infection or severe infectious disease requiring therapy (bacterial, viral or fungal) as per the discretion of the treating physician.
* Presence of another active malignancy (requiring treatment) diagnosed within 12 months with the exception of
* adequately treated non-melanoma skin cancer.
* adequately treated melanoma grade 2 or less.
* cervical intraepithelial neoplasia.
* adequately treated in situ carcinoma of the cervix uteri or carcinoma in situ of breast.
* basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin.
* adequately treated prostate cancer.
* Life-threatening illness with life expectancy < 6 months unrelated to cancer.
* Known HIV positive patients who do not meet the following criteria:
* Cluster of differentiation (CD4) count > 350 cells/mm^3.
* Undetectable viral load.
* Maintained on modern therapeutic regimens utilizing non-cytochrome (CYP)-interactive agents.
* No history of AIDS-defining opportunistic infections.
* Known hepatitis B surface antigen seropositive or known or suspected active hepatitis C infection.

Note: Patients who have isolated positive hepatitis B core antibody (i.e., in the setting of negative hepatitis B surface antigen and negative hepatitis B surface antibody) must have an undetectable hepatitis B viral load. Patients who have positive hepatitis C antibody may be included if they have an undetectable hepatitis C viral load.

* Known hepatic cirrhosis or severe pre-existing hepatic impairment
* Known cardiopulmonary disease defined as:
* Unstable angina.
* Congestive heart failure [New York Heart Association (NYHA) Class III or IV].
* Myocardial infarction (MI) within six months prior to enrollment (subjects who had ischemic heart disease such as a (ACS), MI, and/or revascularization greater than six months before screening and who are without cardiac symptoms may enroll).
* Symptomatic cardiomyopathy.
* Clinically significant pulmonary hypertension requiring pharmacologic therapy.
* Clinically significant arrhythmia.
* History of polymorphic ventricular fibrillation or torsade de pointes.
* Permanent atrial fibrillation [a fib], defined as continuous a fib for ≥ 6 months.
* Persistent a fib, defined as sustained a fib lasting > 7 days and/or requiring cardioversion in the four weeks before screening.
* Grade 3 a fib defined as symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker), or ablation and
* Patients with paroxysmal a fib or < Gr 3 a fib for period of at least six months are permitted to enroll provided that their rate is controlled on a stable regimen.
* Subject has chronic respiratory disease that requires continuous oxygen, or significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, hepatic, cardiovascular disease, or any other medical condition that in the opinion of the investigator would adversely affect his/her participating in this study.
* Treatment with any investigational products, other than the study drugs, within 14 days before the study enrollment or during the study period.
* Uncontrolled high blood pressure (i.e., systolic blood pressure > 180 mm Hg, diastolic blood pressure > 95 mm Hg).
* Prolonged rate corrected QT (QTc) interval ≥ 500 msec, calculated as per institutional guidelines.
* Left ventricular ejection fraction (LVEF) < 50% as assessed by echocardiogram or radionuclide angiography.
* Patients with uncontrolled coagulopathy or bleeding disorder.
* Known moderate-to-severe chronic obstructive pulmonary disease, interstitial lung disease, and pulmonary fibrosis.
* Major surgery within 14 days before the enrollment or a scheduled major surgery during study period.
* Known central nervous system (CNS) involvement with AML.
* Gastrointestinal (GI) tract disease that causes an inability to take oral medications, malabsorption syndrome, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g. Crohn's disease, ulcerative colitis).
* Female subjects who are both lactating and breastfeeding or of childbearing potential who have a positive serum test during screening.
* Female subjects who intend to donate eggs (ova) during the course of this study or four months after receiving their last dose of study drug(s).
* Male subjects who intend to donate sperm during the course of this study or four months after receiving their last dose of study drug(s).
* Has consumed grapefruit, grapefruit products, Seville oranges (including marmalade containing Seville oranges) or star fruit from the day of consent to throughout the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2022-02-27 (Actual)

PRIMARY OUTCOMES:
Recommended phase 2 dose of pevonedistat when co-administered with azacitidine and venetoclax in patients with AML. | Up to 28 days (one cycle) for each dosing cohort.
  The maximum-tolerated dose is defined as the highest dose level at which none of the first three treated subjects, or no more than one of the first six treated subjects, experiences a dose-limiting toxicity.
The toxicity profile of pevonedistat, azacitidine, and venetoclax combination therapy. | Up to 30 days after last dose of study drugs.
  The number of serious adverse events will be measured using NCI-CTCAE v5 criteria.

SECONDARY OUTCOMES:
Complete Remission Rate | Up to five years.
  The number of subjects who achieve complete remission. Complete remission is defined as follows: Bone marrow blasts <5 percent; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0 x 10^9/L (1000/μL); platelet count >100 x 10^9/L (100,000/μL); independence of red cell transfusions.
Complete Remission with Partial Hematological Recovery | Up to five years.
  The number of subjects who achieve complete remission with partial hematological recovery. Complete Remission with Partial Hematological Recovery is defined as:
  Complete remission with partial hematological recovery (CRh) defined as:
  * <5% blasts in the bone marrow.
  * No evidence of disease.
  * Partial recovery of peripheral blood counts.
  * Platelets >50,000/microliter and absolute neutrophil counts >500/microliter.
Partial Remission Marrow | Up to five years.
  The number of subjects who achieve partial remission marrow. Partial Remission Marrow is defined as: Decrease of bone marrow blast percentage to 5 to 15%; and decrease of pretreatment bone marrow blast percentage by at least 50%.
Morphologic Leukemia Free State | Up to five years.
  The number of patients who achieve morphologic leukemia free state. Morphologic Leukemia Free State is defined as: Bone marrow blasts <5%; absence of blasts with Auer rods; absence of extramedullary disease; no hematologic recovery required.
Complete Remission without Minimal Residual Disease | Up to five years.
  The number of patients who achieve CR without minimal residual disease. Complete Remission without Minimal Residual Disease is defined as: CR with negativity for a genetic marker by reverse transcriptase polymerase chain reaction (RT-qPCR), or CR with negativity by MFC.

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Atallah, MD, Principal Investigator — Medical College of Wisconsin
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murthy GSG, Saliba AN, Szabo A, Harrington A, Abedin S, Carlson K, Michaelis L, Runaas L, Baim A, Hinman A, Maldonado-Schmidt S, Venkatachalam A, Flatten KS, Peterson KL, Schneider PA, Litzow M, Kaufmann SH, Atallah E. A phase I study of pevonedistat, azacitidine, and venetoclax in patients with relapsed/refractory acute myeloid leukemia. Haematologica. 2024 Sep 1;109(9):2864-2872. doi: 10.3324/haematol.2024.285014. PMID 38572562